CLINICAL TRIAL: NCT05749523
Title: The Influence of Exercise and Hydration to the Pharmacological Response to Inhaled Terbutalin and Salbutamol in Men
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Insuffient drug supply. Professor Ronald Dahl lefter his position as proffssor in Århus, and all his research were closed.
Sponsor: Vibeke Backer (Other)
Responsible Party: Sponsor-Investigator, Vibeke Backer, Professor, Dr. Med. Chief Physician, Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: 2013-000483-29
Record Dates: First submitted 2013-07-18; First posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Healthy
Keywords: exercise; dehydration; Salbutamol; Terbutalin
MeSH Terms: conditions — Motor Activity; Dehydration | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Exercise (Other): Exercise vs. non-exercise
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Exercise vs non-exercise

SUMMARY:
To investigate the effects of dehydration and exercise for the urine secretion of beta2-agonists.

DETAILED DESCRIPTION:
No studies have examined the influence of factors such as exercise and dehydration on the pharmacokinetic profile of asthmatic drugs (beta2-agonists). Exercise may modify the metabolism and excretion of drugs, and sweat loss during exercise can result in dehydration, both affecting the urine concentration of the drug.

ELIGIBILITY:
Inclusion Criteria:

* men
* aerobic capacity more than 50ml / min / kg
* more than 5h training pr week

Exclusion Criteria:

* smokers
* allergy for the medicine
* chronic diseases

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-11; Primary Completion 2014-04 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Urine concentration of salbutamol and terbutalin | 7 days
  Urine concentration of salbutamol and terbutalin

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke Backer, Professor, Principal Investigator — Dept of Respiratory Medicine, Bispebjerg University Hospital
Locations (1):
- Department of Respiratory Medicine, L, Bispebjerg Hospital,, Copenhagen, NV, Denmark